CLINICAL TRIAL: NCT07117149
Title: Peking University Smart Monitoring and Responsive Technology for Early Childhood Health (PKU-SMART)
Brief Title: Early-Life Strategies for Preventing Obesity in Preschool-aged Children
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: Shandong Maternal and Child Health Hospital (Unknown)
Responsible Party: Principal Investigator, Hai-Jun Wang, Professor in Department of Maternal and Child Health, School of Public Health, Peking University, Peking University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: N0.2025-042
Record Dates: First submitted 2025-08-01; First posted 2025-08-12 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-08

CONDITIONS: Childhood Obesity Prevention
Keywords: Prevention; Intervention; Obesity; Children; Preschool
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Randomization will be performed after the baseline survey. The assessors measuring childrens' health indicators will be blinded at follow-up phases.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- multicomponent intervention (Experimental): This intervention adopts a multi-component, multi-setting approach. Interventions are delivered across kindergartens, families, and healthcare systems, with varying intensity and personalization. Kindergartens serve as the primary implementation site. Trained kindergarten teachers deliver structured health education sessions and conduct regular anthropometric monitoring. Parents play a crucial role in supporting and sustaining children's healthy behaviors. Family-focused components include both health education and behavior change techniques, delivered through offline meetings and the digital health platform. The intervention is supported by a digital health platform ("PKU-SMART Health Platform") where health professionals provide consultation and tailored advice to families. This component aims to reinforce health literacy and access to expert resources.
  Interventions: Behavioral: multicomponent, tiered intervention
- usual-care control (No Intervention): In the control group, participating preschools will receive no intervention during the study period and will continue their routine educational and management practices without modification. After the study is fully completed, control group preschools will have access to all intervention materials and health education resources developed for this project.

INTERVENTIONS:
Behavioral: multicomponent, tiered intervention — Kindergarten: Train teachers and integrate healthy weight management into kindergarten health policies; deliver health education sessions for children; monitor extra dietary intake and physical activity; conduct monthly height and weight measurements.
  Family: Provide multi-format health education (lectures, short videos, articles) to communicate core intervention messages; set health behavior goals and deliver personalized feedback; conduct motivational interviewing in offline parent meetings or by phone.
  Hospital: Offer professional health guidance and medical services. PKU-SMART online platform: Health Education Module; Growth Monitoring Module; Health Behavior Module; Home-Kindergarden Partnership Module.
  Arms: multicomponent intervention

SUMMARY:
The PKU-SMART is a cluster randomized controlled trial conducted in Jinan, Shandong Province, China. This preventive intervention study aims to develop and evaluate a comprehensive obesity intervention framework for preschool children that integrates digital health technologies, multi-sectoral collaboration, and tiered management strategies. The effectiveness and cost-effectiveness of this approach will be assessed.

DETAILED DESCRIPTION:
In the past four decades, the number of children and adolescents with obesity worldwide has increased tenfold, making childhood overweight and obesity one of the most pressing public health issues. In China, the prevalence of overweight and obesity among children under six years old in China has reached 10.4%.

Children with obesity are more likely to develop health problems than their normal-weight peers. The health impacts of childhood obesity often persist into adulthood, significantly increasing the risk of cardiovascular diseases, endocrine and respiratory disorders, cancers, and other chronic conditions. Therefore, the prevention and management of childhood obesity are critical for promoting both immediate and long-term health.

However, current intervention strategies often face challenges such as inconsistent outcomes, poor adherence, and a lack of theoretical foundation. There is a pressing need to develop more effective, scalable, and sustainable approaches.

To address this gap, we propose an intervention(PeKing University Smart Monitoring And Responsive Technology for early childhood health, PKU-SMART), a cluster-randomized preventive trial targeting preschool children. This study will develop and evaluate an innovative, digital health-supported, multi-sector, tiered intervention system aimed at improving preschoolers' health behaviors, reducing obesity prevalence, and supporting long-term weight management.

ELIGIBILITY:
Kindergarten-Level Inclusion Criteria:

* The kindergarten's principal or headmaster consents to participate in the study, and the school demonstrates a high level of cooperation. Required personnel, such as a school health care provider, are available.
* The total number of children in the middle and senior classes (approximately ages 4-6) exceeds 100.
* Teachers and parents of the selected classes demonstrate good compliance and willingness to cooperate with project implementation.

Kindergarten-Level Exclusion Criteria:

* Special kindergartens, such as part-time institutions or schools for children with special needs.
* Kindergartens that have participated or plan to participate in other obesity-related intervention projects within the past year or upcoming year.
* Kindergartens scheduled for closure or relocation within the next two years.

Child-Level Inclusion Criteria:

* The child's primary caregivers can proficiently use smart phones.
* The child is expected to remain enrolled in the same kindergarten for at least one year.
* Parents or legal guardians provide written informed consent for participation.

Child-Level Exclusion Criteria:

* Obesity caused by genetic disorders, endocrine diseases, central nervous system damage, or long-term medication use.
* History of significant diseases affecting major organs such as the heart, lungs, liver, or kidneys (e.g., congenital heart disease, hypertension, asthma).
* Children on special diets, including vegetarianism.
* Children diagnosed with pathological eating disorders or conditions that impair physical activity.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 882 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
children's BMI-Z change | at end of the 9-month intervention
  Calculated based on height and weight using WHO standards. The primary outcome is the difference between two arms in the change of children's BMI-Z scores from baseline to the end of the intervention.

SECONDARY OUTCOMES:
children's BMI-Z change | at 21-month follow-up
  Calculated based on height and weight using WHO standards. The primary outcome is the difference between two arms in the change of children's BMI-Z scores from baseline to the follow-up.
Body Mass Index (BMI) | at the end of the 9-month intervention; at 21-month follow-up.
  BMI is calculated from measured height and weight.
Waist Circumference | at the end of the 9-month intervention; at 21-month follow-up.
  Waist circumference is measured at the midpoint between the lower margin of the last palpable rib and the top of the iliac crest to evaluate central adiposity.
waist-to-Height Ratio, WHtR | at the end of the 9-month intervention; at 21-month follow-up.
  Calculated by dividing waist circumference by height, used as an indicator of fat distribution and risk for metabolic complications.
Systolic and Diastolic Blood Pressures | at the end of the 9-month intervention; at 21-month follow-up.
  Blood pressure is measured using an electronic sphygmomanometer with the child seated after resting, to assess cardiovascular health.
Body Composition | at the end of the 9-month intervention
  Body fat percentage is assessed using a bioelectrical impedance analyzer (MC-780A, TANITA, Tokyo, Japan).
Prevalence and Incidence of Overweight/Obesity | at the end of the 9-month intervention; at 21-month follow-up.
  The proportion of children classified as overweight or obese according to WHO and Chinese standards, including newly identified cases at follow-up.
Children's Eating Behaviors | at the end of the 9-month intervention
  Assessed using the Children's Eating Behavior Questionnaire (CEBQ), measuring dimensions such as food responsiveness, satiety responsiveness, and emotional eating.
Parental Feeding Practices (CPCFBS) | at the end of the 9-month intervention
  Measured using the Chinese Preschooler's Caregivers Feeding Behavior Scale (CPCFBS), evaluating dimensions such as monitoring, pressure to eat, and food restriction.
Time Spent in Physical Activity | at the end of the 9-month intervention
  Evaluated using the Children's Leisure Activities Study Survey (CLASS), assessing the amount and type of physical activity and sedentary behavior, including screen time.
Time Spent in Sedentary Behavior | at the end of the 9-month intervention
  Evaluated using the Children's Leisure Activities Study Survey (CLASS), assessing the amount and type of physical activity and sedentary behavior, including screen time.

CONTACTS AND LOCATIONS:
Overall Officials: Haijun Wang, PhD, Principal Investigator — Peking University
Locations (1):
- Department of Maternal and Child Health, School of Public Health, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared publicly due to ethical considerations. In accordance with the study's ethical approval and informed consent procedures, the data contain potentially sensitive personal health information and are protected to ensure participant confidentiality and privacy. Data access is therefore restricted to authorized research personnel only and cannot be made publicly available.